CLINICAL TRIAL: NCT05741905
Title: Safety and Efficacy of Levofloxacin Combined With Intravenous Thrombolysis for Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LVX-IVT
Record Dates: First submitted 2023-02-06; First posted 2023-02-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Intravenous thrombolysis; Levofloxacin
MeSH Terms: conditions — Ischemic Stroke | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levofloxacin group (Experimental): Levofloxacin 200mg twice per day is administrated.
  Interventions: Drug: Levofloxacin
- Levofloxacin simulant group (Placebo Comparator): Levofloxacin simulant 200mg twice per day is administrated.
  Interventions: Drug: Levofloxacin simulant

INTERVENTIONS:
Drug: Levofloxacin — Levofloxacin is a quinolone antibiotics and newly identified neuro-protective agent. Intravenous thrombolysis is one of the treatments for acute ischemic stroke.
  Other Names: Intravenous Thrombolysis
  Arms: Levofloxacin group
Drug: Levofloxacin simulant — Levofloxacin simulant is placebo. Intravenous thrombolysis is one of the treatments for acute ischemic stroke.
  Other Names: Intravenous Thrombolysis
  Arms: Levofloxacin simulant group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of levofloxacin combined with intravenous thrombolysis in treating acute ischemic stroke

DETAILED DESCRIPTION:
Acute ischemic stroke is a leading cause of disability and mortality. Intravenous thrombolysis is a major therapy for acute ischemic stroke, however, nearly half of patients failed to benefit from it. It is necessary to find new interventions combined to intravenous thrombolysis, which promote the efficacy of intravenous thrombolysis. The investigators' previous studies suggested levofloxacin to be a newly identified neuro-protective agent, which could reduce infarct volume and improve neurologic function in animal models. To evaluate the efficacy and safety of levofloxacin combined with intravenous thrombolysis in treating acute ischemic stroke patients, the prospective, multicenter and randomized controlled trial was designed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. Acute ischemic stroke patients underwent intravenous thrombolysis, treated with ateplase (0.9mg/kg)
3. mRS≤1 before stroke onset, NIHSS ≥ 5 and ≤ 15，la (NIHSS) level of consciousness < 1

Exclusion Criteria:

1. Endovascular treatment
2. Patients using glucocorticoids, antiarrhythmic drugs (class I and class III antiarrhythmic drugs: quinidine, procaine amine, lidocaine, phenytoin sodium, verapamil, etc.), and quinolones within 14 days;
3. Patients with other diseases that may aggravate adverse drug reactions, such as ventricular arrhythmias, prolonged QT interval (male: QTc>430ms, female: QTc>450ms), severe cardiac insufficiency (NYHA functional grade ≥ III), myasthenia gravis, peripheral neuropathy, seizures, tendon-related diseases, severe immune system-related diseases, hematological diseases, active hepatitis or cirrhosis, serious respiratory diseases;
4. Abnormal liver and kidney function: glutamic oxaloacetic transaminase or glutamic pyruvic transaminase exceeds 3 times the upper limit of normal; Direct bilirubin or indirect bilirubin more than 3 times the normal upper limit; Blood creatinine exceeds 1.1 times the upper limit of normal; Creatinine clearance rate≤50ml/min; Urea nitrogen≥ 20mg/dL;
5. Concurrent infection;
6. Fasting blood glucose lower than 3.9 mmol/L;
7. Patients with symptomatic intracranial hemorrhage confirmed by clinical signs and imaging before randomization;
8. Patients allergy to fluoroquinolones or other antibiotics;
9. Patients with a life expectancy less than 3 months or patients unable to complete the study for other reasons;
10. Not willing to be followed up or poor treatment compliance;
11. Patients who are participating in other clinical studies, or have participated in other clinical studies within 3 months before enrollment, or have participated in this study;
12. Other conditions not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
National Institute of Health stroke scale (NIHSS) | in 24 hours of intravenous thrombolysis
  NIHSS ranged from 0 to 42, a low value represents a better outcome
NIHSS at discharge/7 days | discharge/7 days
  NIHSS ranged from 0 to 42, a low value represents a better outcome

SECONDARY OUTCOMES:
Hemorrhagic transformation and symptomatic intracranial hemorrhage | 24h,3 days and discharge/7 days
  defined by computed tomography (CT) brain scan showed bleeding and a concomitant increase in National Institute of Health stroke scale (NIHSS) score of ≥4 points.
Infarct volume after 3 days of Levofloxacin/simulant treatment | Immediately after 3 days of Levofloxacin/simulant treatment
  assessed by magnetic resonance imaging brain scan
Modified rankin scale (mRS) score at 30 days | 30 days
  mRS ranged from 0 to 6, a low value represents a better outcome
mRS score at 90 days | 90 days
  mRS ranged from 0 to 6, a low value represents a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China